| NCT 03403491 | | | |
|---|---|---|---|
| Statistical analyis plan Appendix 1 | date: 26-Jun-2019 | | |
| Protocol | www.clinicaltrials.gov registry no. NCT 03403491 | | |
| Version | 2-Aug-17 | | |
| Amendment 01 | 20-Dec-18 | | |
| Demographic data (for Randomised & Treated dat | • | | |
| Variable | data format | data presentation Statistical comparison | Statistical test used |
| Date of birth | date | descriptive | |
| Age | n (years); calculated (informed consent-date of birth) | descriptive; mean +/- SD, min, max check for treatment order effect (Treated data | set) ? |
| gender | number male/female | frequency, absolute, percentage, histogram check for treatment order effect (Treated data | set) ? |
| ethnicity | number black/white/Asian/other | frequency, absolute, percentage, histogram check for treatment order effect (Treated data | set) ? |
| | number | | |
| primary cause of haemodialysis | glomerular/diabetes/hypertension/hereditary/drug toxicity/other | frequency, absolute, percentage, histogram check for treatment order effect (Treated data | set) ? |
| date 1st ever haemodialysis | date | descriptive | · |
| | n (years); calculated (informed consent-date 1st ever | ····· | |
| time since 1st ever haemodialysis | dialysis) | descriptive; mean +/- SD, min, max check for treatment order effect (Treated data | set) ? |
| usual duration haemodialysis | minutes | descriptive; mean +/- SD, min, max | |
| | number diabetes/hypertension/cardiovascular | | |
| a a markiditi a a | disease/congestive heart failure/peripheral vascular | fraguency check to proportions histogram | not) 2 |
| comorbidities | disease/neurologic/vision impairment/other number permacath/arteriovenous fistula/arteriovenous | frequency, absolute, percentage, histogram check for treatment order effect (Treated data | set) ? |
| vascular access modality | graft/central venous catheter/other | frequency, absolute, percentage, histogram none | |
| usual prescribed haemodialysis sessions/week | number | frequency, absolute, percentage, histogram none | |
| on antihypertensive therapy | number yes/no | frequency, absolute, percentage, histogram check for treatment order effect (Treated data | set) ? |
| number of antihypertensive therapies | number per patient | frequency, absolute, percentage, histogram none | , |
| | number beta-blocker, calcium channel blocker, ACE inhibitor, angiotensin receptor blocker, diuretic, | | |
| classes of antihypertensive | combination, other | frequency, absolute, percentage, histogram none | |
| body mass index | number | descriptive; mean +/- SD, min, max none | |
| Primary endpoint (engagement; Treated dataset) | Level of engagement of patients with patientMpow | , | |
| Variable (in protocol) | data format | data presentation Statistical comparison | Statistical test used |
| patients asked to take part | number | descriptive, count statistical comparison | Statistical lest used |
| · | number | | |
| patients giving informed consent | | p | |
| patients downloading pMp | number | descriptive, count none | |
| patients using pMp at least once | number | descriptive, count none | |
| patients using pMp >once | number | descriptive, count none | |
| frequency of use of pMp | number of days used/number of days in pMp period | descriptive; mean +/- SD, min, max none | |
| date interval informed consent vs. download | number of days | descriptive; mean +/- SD, min, max none | |
| date interval download vs. first use | number of days | descriptive; mean +/- SD, min, max none | |
| requency of use of pMp (any use) | number of days used/number of days in pMp period | descriptive; mean +/- SD, min, max none | |
| requency of weight recorded on pMp | number of days recorded/number of days in pMp period | check for treatment order effect; even balanc randomisation of sequences in >75% adhere descriptive; mean +/- SD, min, max group suggests treatment order effect unlikel | t |
| requency of BP recorded on pMp | number of days recorded/number of days in pMp period | descriptive; mean +/- SD, min, max check for treatment order effect | ? |
| requency of symptoms recorded on pMp | number of days recorded/number of days in pMp period | descriptive; mean +/- SD, min, max none | |
| frequency of fluid intake recorded on pMp | number of days recorded/number of days in pMp period | descriptive; mean +/- SD, min, max none | |

05/03/2020

| patient questionnaire number | number of patients providing response/number of patients starting pMp | descriptive, count | none | |
|---|---|---|---|---|
| patient questionnaire responses | number of responses in each category of 6 questions | descriptive, categorical, count, histogram | none | |
| Secondary endpoints (clinic data) | impact of patientMpower on haemodialysis and sy | mptoms (Treated & >75% adherent datasets) | | |
| /ariable (in protocol) | data format | data presentation | Statistical comparison | Statistical test used |
| proportion of haemodialysis sessions with<br>ultrafiltration rate = 10mL/kg/h</td <td>categorical: number of sessions meeting endpoint/number of sessions</td> <td>count sessions in which endpoint achieved, categorise as yes/no; assign to period</td> <td>run-in vs. active vs. sham within-subject analysis; test for treatment order effect</td> <td>?</td> | categorical: number of sessions meeting endpoint/number of sessions | count sessions in which endpoint achieved, categorise as yes/no; assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| average ultrafiltration rate (mL/kg/h) | number | mean, (all sessions in a period) SD, min, max, assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| average ultrafiltration volume/session (mL) | number | mean, (all sessions in a period) SD, min, max, assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| average ultrafiltration volume/session (mL) | slope of change over time/patient | value vs. time plot, assign to period (graph/patient) | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| proportion of haemodialysis sessions with IDWG =</td <td>categorical: number of sessions meeting endpoint/number of sessions</td> <td>count sessions in which endpoint achieved, categorise as yes/no; assign to period</td> <td>run-in vs. active vs. sham within-subject analysis; test for treatment order effect</td> <td>?</td> | categorical: number of sessions meeting endpoint/number of sessions | count sessions in which endpoint achieved, categorise as yes/no; assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| average IDWG (%) | number | mean, (all sessions in a period) SD, min, max, assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| absolute IDWG (kg) | number | mean, (all sessions in a period) SD, min, max, assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| absolute IDWG (kg) | slope of change over time/patient | value vs. time plot, assign to period (graph/patient) | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | |
| pre-dialysis weight (clinic) | number | mean, (all sessions in a period) SD, min, max, assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| pre-dialysis weight (clinic) | slope of change over time/patient | value vs. time plot, assign to period (graph/patient) | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| post-dialysis weight (clinic) | number | mean, (all sessions in a period) SD, min, max, assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| post-dialysis weight (clinic) | slope of change over time/patient | value vs. time plot, assign to period (graph/patient) | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| pre-dialysis SBP (clinic) | number | mean, (all sessions in a period) SD, min, max, assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| pre-dialysis DBP (clinic) | number | mean, (all sessions in a period) SD, min, max, assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| pre-dialysis SBP (clinic) | slope of change over time/patient | value vs. time plot, assign to period (graph/patient) | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| pre-dialysis DBP (clinic) | slope of change over time/patient | value vs. time plot, assign to period (graph/patient) | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| post-dialysis SBP (clinic) | number | mean, (all sessions in a period) SD, min, max, assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| post-dialysis DBP (clinic) | number | mean, (all sessions in a period) SD, min, max, assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| post-dialysis SBP (clinic) | slope of change over time/patient | value vs. time plot, assign to period (graph/patient) | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| post-dialysis DBP (clinic) | slope of change over time/patient | value vs. time plot, assign to period (graph/patient) | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| medication adherence | number of days adherence reported/number of days in pMp period | count, mean, SD, min, max | none | |
| inplanned haemodialysis sessions | number of unplanned sessions | count, allocate to period: run-in, sham or pMp | none | |
| clinic dry weight [pre-dialysis weight (kg) -ultrafiltration goal volume (L)] | number | mean, (all sessions in a period) SD, min, max, assign to period | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| clinic dry weight [pre-dialysis weight (kg) -ultrafiltration goal volume (L)] | slope of change over time/patient | value vs. time plot, assign to period (graph/patient) | run-in vs. active vs. sham within-subject analysis; test for treatment order effect | ? |
| Secondary endpoints (patient-reported data) | impact of patientMpower on haemodialysis and sy | mptoms (Treated dataset) | | |
| Variable (in protocol) | data presentation | | Statistical comparison | |

05/03/2020 2

| symptoms (any reported) on >/= one day | number of patients reporting any symptom >/=once | descriptive, count | none | |
|---|---|---|---|---|
| nax number of symptoms reported on >/= one day | number of patients reporting 0, 1, 2, 3, 4, 5 or 6 symptoms on >/= one day | descriptive, categorical, count, histogram | none | |
| ymptoms (muscle cramp) reported on >/= one day | number of patients reporting this symptom >/= once | descriptive, count | none | |
| symptoms (muscle cramp) worst severity | number of patients reporting this symptom none, 1-2, 3-4 or >4 times/day >/= once | descriptive, categorical, count, histogram | none | |
| symptoms (muscle cramp) severity over time | Assign severity score to symptom (not at all =0, 1,2 /d= 1, 2-4/d = 2, >4/d =3); trend over time | value vs. time plot (graph/patient) | none | |
| symptoms (feeling washed out) reported on >/= one day | number of patients reporting this symptom >/= once | descriptive, count | none | |
| symptoms (feeling washed out) worst severity | number of patients reporting this symptom none, mild, moderate, severe >/= once | descriptive, categorical, count, histogram | none | |
| symptoms (feeling washed out) severity over time | Assign severity score to symptom (not at all =0, mild = 1, moderate = 2, severe =3); trend over time | value vs. time plot (graph/patient) | none | |
| symptoms (light-headedness) reported on >/= one day | number of patients reporting this symptom >/= once | descriptive, count | none | |
| symptoms (light-headedness) worst severity | number of patients reporting this symptom none, mild, moderate, severe >/= once | descriptive, categorical, count, histogram | none | |
| symptoms (light-headedness) over time | Assign severity score to symptom (not at all =0, mild = 1, moderate = 2, severe =3); trend over time | value vs. time plot (graph/patient) | none | |
| symptoms (shortness of breath) reported on >/= one day | number of patients reporting this symptom >/= once | descriptive, count | none | |
| symptoms (shortness of breath) worst severity | number of patients reporting this symptom none, mild, moderate, severe >/= once | descriptive, categorical, count, histogram | none | |
| symptoms (shortness of breath) severity over time | Assign severity score to symptom (not at all =0, mild = 1, moderate = 2, severe =3); trend over time | value vs. time plot (graph/patient) | none | |
| symptoms (swollen ankles) reported on >/= one day | number of patients reporting this symptom >/= once | descriptive, count | none | |
| symptoms (swollen ankles) worst severity | number of patients reporting this symptom none, mild, moderate, severe >/= once | descriptive, categorical, count, histogram | none | |
| symptoms (swollen ankles) severity over time | Assign severity score to symptom (not at all =0, mild = 1, moderate = 2, severe =3); trend over time | value vs. time plot (graph/patient) | none | |
| symptoms (cough) reported on >/= one day | number of patients reporting this symptom >/= once | descriptive, count | none | |
| luid intake reported on >/= one day | number of patients reporting fluid intake >/= once | descriptive, count | none | |
| maximum fluid intake | number of patients reporting small, medium or large fluid intake >/= once | descriptive, categorical, count, histogram | none | |
| luid intake quantity over time | Assign score to amount (small =1, medium = 2, large =3); trend over time | value vs. time plot (graph/patient) | none | |
| Farget weight | slope of change over time/patient | descriptive; value vs. time plot (target weight is as entered on pMp), graph/patient | none | |
| Farget weight/dry weight | slope of change over time/patient | descriptive; value vs. time plot (target weight is as entered on pMp; dry weight from haemodialysis clinic data); graph/patient | none | |
| veight change vs. target weight | number of times in 0.00-1.99%, 2.00-3.49%, 3.50-4.49% and >/=4.5% gain vs. target per patient (positive or negative) | descriptive, categorical, count, histogram (graph/patient & total patient population) | none | |
| weight change vs. target weight | slope of change over time/patient | descriptive; value vs. time plot (target weight is as entered on pMp), graph/patient | none | |
| SBP (seated) | number | descriptive, mean, SD, min, max of all values (per patient) | none | |
| SBP (seated) | slope of change over time/patient | descriptive; value vs. time plot, graph/patient | none | |
| DBP (seated) | number | descriptive, mean, SD, min, max of all values (per patient) | none | |
| DBP (seated) | slope of change over time/patient | descriptive; value vs. time plot, graph/patient | none | |
| nferior vena cava data | variable | data format | Statistical comparison | Statistical test used |
| | | descriptive, count, mean, SD, min, max; allocate to period (run-in, sham, active) | | |
| ongitudinal diameter (mm) | number | active) | | |

05/03/2020 3

## 20190626 Statistics analysis plan Appendix 1

| longitudinal diameter (mm) | slope of change over time/patient | value assigned to period (run-in, active, sham); graph/patient | run-in vs. active vs. sham within-subject<br>analysis; test for treatment order effect; if none<br>compare mean total population values per<br>period | ? |
|---|---|---|---|---|
| transverse diameter (mm) | slope of change over time/patient | value assigned to period (run-in, active, sham); graph/patient | run-in vs. active vs. sham within-subject<br>analysis; test for treatment order effect; if none<br>compare mean total population values per<br>period | ? |
| Collapsibility | 50% collapsible on inspiration? | descriptive, categorical, count | run-in vs. active vs. sham within-subject<br>analysis; test for treatment order effect; if none<br>compare mean total population values per<br>period | |

05/03/2020 4